CLINICAL TRIAL: NCT04504357
Title: Integrating U=U Into HIV Counseling in South Africa
Acronym: INTUIT-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-40706; R34MH122323 (NIH)
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: Antiretroviral treatment (ART); Person living with HIV (PLWH); Treatment-as-prevention (TasP); Undetectable=Untransmittable (U=U); HIV counseling; South Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A- No intervention (No Intervention): Participants randomized to Arm A received no research intervention.
- Arm B- "Undetectable & You" App (Experimental): Participants randomized to Arm B interacted with "Undetectable & You" a tablet-based treatment literacy App that shared the science of U=U through testimonials of PLHIV and their partners. Participants in Arm B also received monthly text messages related to the themes of the App.
  Interventions: Behavioral: Tablet based U=U app; Other: Text messages

INTERVENTIONS:
Behavioral: Tablet based U=U app — Tablet based "app" focusing on TasP/U=U videos on: a) the science of TasP/U=U including risks, (b) benefits to self (e.g. psychological benefits, ability to have children), (c) benefits to partners (e.g. secondary prevention), (d) benefits to society (e.g. AIDS-free generation), and (e) TasP self-efficacy, including viral load (VL) literacy, disclosure, and couples testing.
  Arms: Arm B- "Undetectable & You" App
Other: Text messages — Monthly text messages reinforcing intervention content
  Arms: Arm B- "Undetectable & You" App

SUMMARY:
The near-elimination of HIV transmission with antiretroviral therapy (ART) has provided the world with a clear path to end the HIV epidemic through the mass provision of ART at diagnosis, i.e. test-and-treat. Despite the substantial prevention benefits of ART, the investigators found minimal knowledge of treatment-as-prevention (TasP) in two population-based surveys recently conducted in South Africa. In addition, current public health messaging and clinical HIV counselling in South Africa do not emphasize the prevention benefits of ART.

In this formative research study the investigators developed an app-based educational video intervention that provides information on Undetectable = Untransmittable (U=U) that is locally-appropriate and can be integrated into routine HIV counselling. The intervention was be piloted in a clinical trial of patients in South Africa receiving HIV post-test and adherence counselling services, to determine feasibility and acceptability, impact on U=U knowledge and attitudes, impact on stigma and psychological well being, and preliminary evidence for ART uptake and adherence.

The study builds on a longstanding collaboration between Boston University and the Health Economics and Epidemiology Research Office (HE2RO) at the University of Witwatersrand in Johannesburg, South Africa. The study is highly innovative because the investigators take a novel approach - disseminating information on the prevention benefits of ART - to improve the wellbeing of people living with HIV (PLWH) and motivate early uptake of ART in South Africa.

The investigators hypothesized that disseminating information about U=U and treatment-as-prevention could increase ART adherence, retention, and viral suppression, enabling countries to maximize the impact of test-and-treat.

DETAILED DESCRIPTION:
We developed a U=U-focused HIV treatment literacy App called "Undetectable & You", to integrate U=U into HIV counseling in South Africa. We then piloted the App in a randomized clinical trial.

The randomized pilot trial was conducted at three public sector clinics in Johannesburg, South Africa, to establish intervention acceptability, effects on knowledge and attitudes, and preliminary impact on ART uptake, adherence, retention, and viral suppression (n=135).

Patients completing HIV post-test or adherence counseling were referred to study staff and randomized 1:1 to no intervention (Arm A) vs. a ~20min interaction with "Undetectable & You", a tablet-based App developed to disseminate information about U=U via PLHIV testimonials (Arm B). Participants in Arm B also received monthly text messages reinforcing intervention content. The order of the messages was randomized to ascertain whether different messages were better at driving engagement with the App.

Investigators assessed feasibility and acceptability of the "Undetectable & You" App, resonance of different key messages and videos in the App, and its impact on knowledge and attitudes related to TasP. Additionally, ART uptake, appointment adherence, retention on treatment, and viral monitoring were assessed in clinical records through six months, with VL data collected through 10 months. Qualitative exit interviews were conducted with participants and clinic staff (n=30).

In addition to the primary and secondary outcomes specified below, we assessed for effect modification in the primary outcome of viral suppression by key constructs of our theoretical model and participant demographics.

ELIGIBILITY:
Inclusion Criteria:

* receiving HIV care at a public sector health facility in South Africa
* Speaks English, Zulu, or Sotho

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bor, ScD SM, Principal Investigator — BU School of Public Health, Global Health
Locations (3):
- South Africa (3):
  - Primary Health Clinic A, Johannesburg, Gauteng
  - Primary Health Clinic B, Johannesburg, Gauteng
  - Primary Health Clinic C, Johannesburg

IPD SHARING:
Plan to Share IPD: Yes
Replication data, code, and protocol (including SAP) will be posted on a public repository when the trial results manuscript is published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At manuscript publication.
Access Criteria: Publicly accessible

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 135 participants were enrolled and prior to randomization, 4 participants exited the study (2 during the baseline survey and 2 who did not have clinical charts) leaving 131 to be randomized into the two study arms. 67 participants were randomized into Arm A/No intervention and 64 were randomized into Arm B/"Undetectable & You" app.
Period: Wave 1 Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Started | 67 | 64
Completed | 67 | 64
Not Completed | 0 | 0
Period: Wave 2 Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 64 | 131
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 43 | 33 | 76
  Male | 24 | 30 | 54
  Neither male nor female | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 67 | 64 | 131

OUTCOME MEASURES:

1. Primary Outcome: Documented HIV Viral Load <200 Copies/mL at 3-10 Months
Description: As documented in linked clinical records. The first viral load (VL) value taken during the period 3-10 months after baseline. Outcome will be defined as documented viral suppression among all patients: 1 = VL<200; 0 = VL>=200 OR no documented VL. The 200 copy threshold matches WHO definition for "zero transmission risk".
Time Frame: 3-10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 22 | 33

2. Secondary Outcome: Started ART Within 30 Days of Baseline
Description: As documented in linked clinical records
Time Frame: 0-1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 64 | 64

3. Secondary Outcome: ART Refills Beyond 30 Days
Description: Any ART refills recorded in clinical records after 30 days post-enrollment.
Time Frame: 1-6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 55 | 60

4. Secondary Outcome: ART Uptake and First Refill Within 60 Days (Composite Outcome)
Description: Indicator = 1 if the participant started ART and returned to the clinic for their first ART medication refill within 60 days after enrollment. Indicator = 0 if the participant did not start ART, or if patient started ART but did not have a medication refill within 60 days of enrollment.
Time Frame: 0-2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 50 | 53

5. Secondary Outcome: Retained in Care at 1-2 Months
Description: Any ART refills during months 1-2 post enrollment.
Time Frame: 1-2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 54 | 55

6. Secondary Outcome: Retained in Care at 3-4 Months
Description: Any ART refills during months 3-4 post enrollment.
Time Frame: 3-4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 48 | 54

7. Secondary Outcome: Retained in Care at 5-6 Months
Description: Any ART refills during months 5-6 post enrollment.
Time Frame: 5-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 38 | 47

8. Secondary Outcome: Viral Load Monitoring at 3-10 Months
Description: Based on linked clinical records, 3-10 months after baseline
Time Frame: 3-10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 67 | 64
Participants | 30 | 40

9. Secondary Outcome: Mean Percent Perceived Transmission Risk When PLHIV is on ART and Virally Suppressed
Description: Likelihood of HIV transmission (on a 0 to 100 scale) in a hypothetical mixed-status couple after a year of weekly condomless sex, where the HIV+ partner is on ART. Higher scores are associated with higher perceived risk.
Time Frame: after intervention (on average 6 months)
Population: Only wave 2 participants (34 in Arm A and 34 in Arm B) were assessed for this outcome measure.
Measure: Number; unit: percentage of perceived risk
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
Number analyzed (Participants) | 34 | 34
percentage of perceived risk | 37.7 | 12.7

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Arm A- No Intervention | Arm B- "Undetectable & You" App
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT04504357/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT04504357/ICF_000.pdf